CLINICAL TRIAL: NCT03050697
Title: A Prospective, Multicenter Study to Evaluate the Safety and Performance of the Exchangeable ClarVista HARMONI Modular Toric Intraocular Lens System for the Treatment of Pre-Existing Corneal Astigmatism and Aphakia Following Cataract Surgery
Brief Title: Evaluation of the Safety and Performance of the HARMONI® Toric Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ClarVista Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-00004
Record Dates: First submitted 2016-09-14; First posted 2017-02-13 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Aphakia; Corneal Astigmatism; Cataract
Keywords: Toric; Intraocular lens
MeSH Terms: conditions — Aphakia; Astigmatism; Cataract | interventions — Cataract Extraction; Lenses, Intraocular; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- HMTIOL (Experimental): HARMONI® Modular Toric Intraocular Lens implanted in the capsular bag following removal of the cataractous lens, intended for lifetime use
  Interventions: Device: HARMONI® Modular Toric Intraocular Lens; Procedure: Cataract extraction with intraocular lens (IOL) implantation

INTERVENTIONS:
Device: HARMONI® Modular Toric Intraocular Lens — Two-component system consisting of a base and a separate toric optic
  Other Names: HMTIOL
Procedure: Cataract extraction with intraocular lens (IOL) implantation — Cataract removal via manual phacoemulsification, followed by HMTIOL implantation

SUMMARY:
The purpose of this study was to evaluate the safety and effectiveness of the HARMONI® Modular Intraocular Lens System with a toric optic (HMTIOL) in subjects with pre-existing corneal astigmatism in need of cataract surgery.

DETAILED DESCRIPTION:
Subjects with visually significant bilateral cataracts (cortical, nuclear, posterior subcapsular, or a combination) were implanted unilaterally (in one eye only) or bilaterally (in both eyes) with the HMTIOL. A total of 7 study visits were planned, including a preoperative visit, operative visits for each eye, and 4 follow-up visits at 1 day, 1 week, 1 month, and 3 months postoperative. The total duration of participation for each subject was up to 6 months, including the preoperative period (up to 3 months).

Alcon Research, LLC, acquired ClarVista Medical in 2017. This study was designed and conducted by ClarVista Medical, Inc. The study results were collected, analyzed, and provided by ClarVista Medical, Inc. to Alcon Research, LLC.

ELIGIBILITY:
Key Inclusion Criteria:

* Planned removal of visually significant bilateral cataract by manual phacoemulsification cataract extraction
* Pre-existing corneal astigmatism in at least 1 eye of 0.75 to 2.50 diopter (D)
* Target dioptric lens power within the range of 16 - 26 D
* Willing to discontinue contact lens wear for the duration of the study
* BCVA projected to be ≤0.2 logarithm minimum angle of resolution (LogMAR)
* Stable cornea
* Dilated pupil size at least 7.0 millimeters (mm)
* Able to understand and provide informed consent.

Key Exclusion Criteria:

* History of any intraocular or corneal surgery in study eye (including refractive)
* Pregnant or lactating
* History of any clinically significant retinal pathology or ocular diagnosis in study eye that could alter or limit final postoperative visual prognosis
* History of ocular conditions which could affect the stability of the IOL in study eye
* Any anterior segment pathology likely to increase the risk of complications from phacoemulsification cataract extraction in study eye
* Any visually significant intraocular media opacity other than cataract in study eye
* Uncontrolled glaucoma in study eye
* Uncontrolled systemic disease
* Severe dry eye that would impair the ability to obtain reliable study measurements
* Systemic medication that may confound the outcome or increase the intraoperative and postoperative risk to the subject.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Surgical, Study Director — Alcon Research, LLC
Locations (1):
- ClarVista Investigative Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one investigative site located in New Zealand.
Pre-assignment Details: Of the 16 subjects (25 eyes) enrolled in the study, 4 subjects (7 eyes) were exited prior to implantation as screen failures, and 1 eye in 1 subject was exited prior to implantation due to a medical condition. This reporting group includes all implanted subjects (12) and eyes (17).
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | HMTIOL
Started | 12; 17 eyes
Completed | 12; 17 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: All Implanted Subjects
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0
  Black | 0
  Caucasian | 10
  Other | 2
Region of Enrollment [Number; unit: participants]
  New Zealand | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Manifest Refraction Cylinder (MRCYL) for Eyes Implanted With HMTIOL
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. Manifest refraction cylinder is the amount of added correction needed to compensate for any astigmatism that may be present. MRCYL was measured in diopters and reported as a negative number, with a less negative number indicating a lesser amount of added correction. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Number analyzed (eyes) | 17
diopter
  Month 1 postoperative | -0.50 (0.95)
  Month 3 postoperative | -0.57 (0.98)

2. Primary Outcome: Mean Manifest Refraction Cylinder (MRCYL) Prediction Error (PE) for Eyes Implanted With HMTIOL
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. Manifest refraction cylinder is the amount of power needed to correct any astigmatism that may be present. MRCYL was measured in diopters and reported as a negative number. MRCYL PE was calculated as postoperative MRCYL adjusted to 6 meters minus MRCYL target residual refractive error (TRRE), with a lower absolute value indicating a more accurate cylinder power calculation. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Number analyzed (eyes) | 17
diopter
  Month 1 postoperative | 0.01 (0.26)
  Month 3 postoperative | -0.03 (0.29)

3. Primary Outcome: MRCYL PE for Eyes Implanted With HMTIOL Per Vector Analyses
Description: Manifest refraction cylinder is the amount of power needed to correct any astigmatism that may be present. MRCYL PE is calculated as postoperative MRCYL adjusted to 6 meters minus MRCYL target residual refractive error (TRRE), with a lower absolute value indicating a more accurate cylinder power calculation. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative
Population: Vector analyses (Eydelman 2006) based on the cylinder power and axis were planned but were not performed.
Arm/Group | HMTIOL
Number analyzed (Participants) | 0

4. Primary Outcome: Mean Reduction in Cylinder Power for Eyes Implanted With HMTIOL
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. Manifest refraction cylinder is the amount of power needed to correct any astigmatism that may be present. MRCYL was measured in diopters and reported as a negative number. Cylinder power reduction was calculated as the absolute preoperative magnitude of corneal cylinder (K) minus the absolute postoperative magnitude of MRCYL at the corneal plane. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 preoperative), Month 3 postoperative
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Number analyzed (eyes) | 17
diopter | 1.15 (0.63)

5. Primary Outcome: Mean Percent Reduction in Cylinder Power for Eyes Implanted With HMTIOL
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. Manifest refraction cylinder is the amount of power needed to correct any astigmatism that may be present. MRCYL was measured in diopters and reported as a negative number. Cylinder power reduction was calculated as the absolute preoperative magnitude of corneal cylinder (K) minus the absolute postoperative magnitude of MRCYL at the corneal plane. Therefore, the cylindrical power percent reduction was the cylinder power reduction divided by the absolute value of preoperative magnitude of corneal cylinder (K) × 100. A higher number (greater percent reduction) indicates better astigmatism correction by the toric IOL. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 preoperative), Month 3 postoperative
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit
Measure: Mean (Standard Deviation); unit: percent reduction
Units Other Than Participants: eyes
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Number analyzed (eyes) | 17
percent reduction | 76.2 (27.4)

6. Primary Outcome: Mean Manifest Refraction Spherical Equivalent (MRSE) Prediction Error (PE)
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. The manifest refraction spherical equivalent (MRSE) was calculated as follows: sphere + 1/2 cylinder, and measured in diopters (D). MRSE PE was calculated as postoperative MRSE adjusted to 6 meters minus MRSE target residual refractive error (TRRE). The lower the absolute number, the more accurate the IOL power calculation is. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Number analyzed (eyes) | 17
diopter
  Month 1 postoperative | 0.14 (0.41)
  Month 3 postoperative | 0.26 (0.43)

7. Primary Outcome: Mean Absolute Misalignment of IOL Meridian - Target Versus Actual at Operative Visit
Description: Absolute misalignment of IOL meridian was defined as the summation of IOL misplacement and IOL rotation. A lower number indicates minimal IOL misalignment. No formal statistical hypothesis testing was planned.
Time Frame: Day 0 (operative)
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Number analyzed (eyes) | 17
degrees | 2.6 (1.7)

8. Primary Outcome: Mean Absolute Rotation of IOL Meridian by Visit
Description: IOL orientation was measured with slit-lamp photography. IOL rotation was defined as the difference between axis of IOL orientation on the day of surgery and the subsequent postoperative visit. IOL rotation was measured in degrees. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 preoperative), Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Groups:
- HMTIOL - Day 1 Postoperative: HARMONI® Modular Toric Intraocular Lens implanted in the capsular bag following removal of the cataractous lens, intended for lifetime use
Arm/Group | HMTIOL - Day 1 Postoperative
Number analyzed (Participants) | 12
Number analyzed (eyes) | 13
degrees
  Rotation from operative to Day 1 postoperative | 1.9 (1.8)
  Rotation from operative to Week 1 postoperative | 2.3 (1.6)
  Rotation from operative to Month 1 postoperative | 2.9 (2.2)
  Rotation from operative to Month 3 postoperative | 2.4 (2.3)

9. Primary Outcome: Number of Eyes With Absolute Rotation of IOL Meridian by Visit
Description: IOL orientation was measured with slit-lamp photography. IOL rotation was defined as the difference between axis of IOL orientation on the day of surgery and the subsequent postoperative visit. IOL rotation was measured in degrees and is reported categorically. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 preoperative), Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit. Analysis of IOL rotation was planned for rotation categories of ≤ 5°, < 10°, < 20°, and < 30°. Instead, IOL rotation was reported for categories of ≤ 5°, > 5° to ≤ 10°, > 10° to ≤ 20°, and > 20°.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- HMTIOL - Week 1 Postoperative; HMTIOL - Month 1 Postoperative; HMTIOL - Month 3 Postoperative: HARMONI® Modular Toric Intraocular Lens implanted in the capsular bag following removal of the cataractous lens, intended for lifetime use
Arm/Group | HMTIOL - Day 1 Postoperative | HMTIOL - Week 1 Postoperative | HMTIOL - Month 1 Postoperative | HMTIOL - Month 3 Postoperative
Number analyzed (Participants) | 12 | 12 | 12 | 12
Number analyzed (eyes) | 13 | 13 | 13 | 13
eyes
  Rotation from operative ≤ 5 degrees | 12 | 12 | 12 | 12
  Rotation from operative > 5 to ≤ 10 degrees | 1 | 1 | 1 | 1
  Rotation from operative > 10 to ≤ 20 degrees | 0 | 0 | 0 | 0
  Rotation from operative > 20 degrees | 0 | 0 | 0 | 0

10. Primary Outcome: Percentage of Eyes With Best Corrected Distance Visual Acuity (BCDVA) by Visit
Description: Visual Acuity of the eye was tested while reading charts at 20-foot equivalent distance from the participant with the correction obtained from manifest refraction testing. BCDVA is reported categorically using the Snellen fraction, which compares the participant's result to the result expected from a 'normal' visual system. The numerator represents the distance between the participant and the chart, and the denominator represents the distance at which a person with 'normal' vision would be able to discern the same letter size. 20/20 is considered to be 'normal' vision, whereas visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. A larger denominator, therefore, indicates a lower visual acuity. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 preoperative), Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- HMTIOL - Baseline (Day 0 Preoperative); HMTIOL - Week 1 Postoperative; HMTIOL - Month 1 Postoperative; HMTIOL - Month 3 Postoperative: HARMONI® Modular Toric Intraocular Lens implanted in the capsular bag following removal of the cataractous lens, intended for lifetime use
Arm/Group | HMTIOL - Baseline (Day 0 Preoperative) | HMTIOL - Week 1 Postoperative | HMTIOL - Month 1 Postoperative | HMTIOL - Month 3 Postoperative
Number analyzed (Participants) | 12 | 12 | 12 | 12
Number analyzed (eyes) | 17 | 17 | 17 | 17
percentage of eyes
  20/20 Snellen or Better | 35.3 | 82.4 | 82.4 | 88.2
  20/25 Snellen or Better | 47.1 | 88.2 | 94.1 | 88.2
  20/32 Snellen or Better | 64.7 | 88.2 | 94.1 | 100.0
  20/40 Snellen or Better | 64.7 | 94.1 | 94.1 | 100.0
  Worse than 20/40 Snellen | 35.3 | 5.9 | 5.9 | 0.0

11. Primary Outcome: Percentage of Eyes With Uncorrected Distance Visual Acuity (UCDVA) by Visit
Description: Visual Acuity of the eye was tested while reading charts at 20-foot equivalent distance from the participant with an optical infinity adjustment of +0.25 diopter (D). UCDVA is reported categorically using the Snellen fraction, which compares the participant's result to the result expected from a 'normal' visual system. The numerator represents the distance between the participant and the chart, and the denominator represents the distance at which a person with 'normal' vision would be able to discern the same letter size. 20/20 is considered to be 'normal' vision, whereas visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. A larger denominator, therefore, indicates a lower visual acuity. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 preoperative), Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye: All eyes with successful HMTIOL implantation and data at visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | HMTIOL - Baseline (Day 0 Preoperative) | HMTIOL - Day 1 Postoperative | HMTIOL - Week 1 Postoperative | HMTIOL - Month 1 Postoperative | HMTIOL - Month 3 Postoperative
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Number analyzed (eyes) | 17 | 17 | 17 | 17 | 17
percentage of eyes
  20/20 Snellen or Better | 0.0 | 23.5 | 52.9 | 47.1 | 52.9
  20/25 Snellen or Better | 5.9 | 35.3 | 76.5 | 70.6 | 76.5
  20/32 Snellen or Better | 35.3 | 70.6 | 76.5 | 76.5 | 76.5
  20/40 Snellen or Better | 47.1 | 82.4 | 88.2 | 88.2 | 88.2
  Worse than 20/40 Snellen | 52.9 | 17.6 | 11.8 | 11.8 | 11.8

12. Primary Outcome: Standard Error of the Mean in Lens Power A-constant for Refinement
Description: The A-constant (lens power constant) is a theoretical value that is used to calculate the power of the intraocular lens. It relates the lens power to the eye's axial length and keratometry. It is not expressed in units; it is specific to the design of the IOL and its intended location and orientation within the eye.
  A-constants are typically empirically developed for new IOLs based on hundreds of clinical uses. Data from a sufficient number of eyes are needed in order to reduce bias due to surgical technique, unusual eyes, and differences in equipment, such that the standard error of the mean in the lens power constant would be less than ±0.10 mm (approximately ±0.2 diopter). This study represented the first clinical use of the HMTIOL.
Time Frame: Day 0 operative
Population: The planned sample size of 200 eyes was calculated based on the planned refinement of the A-Constant; however, due to the change in the study design, a sample size of 30 was targeted and a total of 17 eyes were implanted. Refinement of the A-Constant was planned, but not completed, due to the change in study design. No data was collected.
Arm/Group | HMTIOL
Number analyzed (Participants) | 0

13. Primary Outcome: Number of Ocular Adverse Events Through Month 3
Description: Ocular adverse events were identified as outlined in ISO 11979-2014 Annex B. No formal statistical hypothesis testing was planned.
Time Frame: Up to Month 3 postoperative
Population: Safety Analysis: All eyes with attempted study lens implantation (successful or aborted after contact with the eye)
Measure: Number; unit: event
Units Other Than Participants: eyes
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Number analyzed (eyes) | 17
event
  Astigmatism | 1
  Ciliary zonular dehiscence | 1
  Intraocular injection | 1
  Macular oedema | 1
  Vitrectomy | 1

14. Primary Outcome: Number of Device-Related Secondary Surgical Interventions (SSI) Other Than Optic Exchange and Rotational Adjustment of the HMTIOL
Description: A secondary surgical intervention (SSI) was defined as a surgical procedure that occurred after primary implantation and was conducted for the purpose of resolving residual refractive error (RRE) and optimizing visual outcomes. No formal statistical hypothesis testing was planned.
Time Frame: Up to Month 3 postoperative
Population: Safety Analysis: All eyes with attempted study lens implantation (successful or aborted after contact with the eye)
Measure: Number; unit: SSI
Units Other Than Participants: eyes
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Number analyzed (eyes) | 17
SSI | 1

15. Primary Outcome: Number of Device Deficiencies Post Implantation
Description: A device deficiency was defined as a failure of the device to meet its performance specifications or expectations, or otherwise not perform as intended. This could include either a malfunction or damage to the device or any part thereof, regardless of the source of malfunction or damage, including user error, and regardless of the presence of injury (or lack thereof) to subject, user, or bystander. No formal statistical hypothesis testing was planned.
Time Frame: Up to Month 3 postoperative
Population: Safety Analysis: All eyes with attempted study lens implantation (successful or aborted after contact with the eye)
Measure: Number; unit: device deficiency
Units Other Than Participants: eyes
Arm/Group | HMTIOL
Number analyzed (Participants) | 12
Number analyzed (eyes) | 17
device deficiency | 0

16. Primary Outcome: Number of Eyes With Preservation of Best Corrected Distance Visual Acuity (BCDVA) at Month 1 and Month 3
Description: Preservation of BCDVA was defined in terms of lines lost when reading the ETDRS chart at each visit compared to the prior best-achieved BCDVA. Loss of < 1 line included subjects with less than a 1 line loss, no change or improvement in BCDVA. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative
Population: Safety Analysis: All eyes with attempted study lens implantation (successful or aborted after contact with the eye)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | HMTIOL - Month 1 Postoperative | HMTIOL - Month 3 Postoperative
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 17 | 17
eyes
  Loss < 1 line | 16 | 16
  Loss >= 1 line | 1 | 1
  Loss >= 2 lines | 0 | 0
  Loss >= 3 lines | 0 | 0
  Loss >= 4 lines | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent until study exit (up to 6 months).
Description: An adverse event was defined as any untoward medical event that does not necessarily have a causal relationship to the study device or protocol. "At Risk" population for ocular adverse events is reported with unit of eye.
Groups:
- HMTIOL - Nonocular AEs: All subjects with attempted study lens implantation (successful or aborted after contact with the eye)
- HMTIOL - Ocular AEs: All eyes with attempted study lens implantation (successful or aborted after contact with the eye)
Arm/Group | HMTIOL - Nonocular AEs | HMTIOL - Ocular AEs
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 0/12 | 2/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HMTIOL - Nonocular AEs (N=12) | HMTIOL - Ocular AEs (N=17)
Astigmatism (Eye disorders) | 0 | 1
Macular oedema (Eye disorders) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 — Recorded as ciliary zonular dehiscence in Outcome Measure 13
Intra-ocular injection (Surgical and medical procedures) | 0 | 1
Vitrectomy (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT03050697/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT03050697/SAP_001.pdf